CLINICAL TRIAL: NCT02660892
Title: Determination of Threonine Requirements and the Metabolic Availability of Threonine From Food Sources in Healthy School-aged Children
Brief Title: Determination of Threonine Requirements in Healthy School-aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H15-02691
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Threonine Requirements in Children
Keywords: IAAO; Threonine; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Protein Intake (Experimental): Threonine intake - Dietary supplement
  Interventions: Dietary Supplement: Protein intake

INTERVENTIONS:
Dietary Supplement: Protein intake — Oral consumption of eight hourly experimental meals
  * 4 tracer free experimental meals containing a mixture of free amino acids and calories from protein free flavoured liquid, protein free cookies and corn oil
  * 4 isotopically labeled experimental meals.

SUMMARY:
Threonine is an indispensable amino acid (nutrient containing nitrogen), which cannot be made in the body and must be consumed from food. Amino acids are the building blocks of protein in your body, and need to be eaten in required amounts to maintain health and growth. Deficiency in threonine can affect small intestine growth due to its structural importance in the intestinal protein mucin. While threonine is found in many foods, deficiency can occur in developing countries where nutrition is primarily plant based, and low in available protein.

Therefore, the purpose of this study is to determine the requirement of the indispensable amino acid Threonine, in school-aged children (6-10y). Secondly, we wish to determine the availability of threonine from three test proteins (soy, green pea, casein).

DETAILED DESCRIPTION:
The threonine intake requirement for children are based on factorial calculations. In the current study we will use a new and modern technique, the indicator amino acid oxidation technique (IAAO), to determine threonine requirements in children.

This technique is a newer technique which involves the consumption of protein shakes composed of specific amounts of threonine mixed with a stable isotope tracer. The oxidation of this isotope will be measured in urine and breath to determine a breakpoint (requirement) of threonine.

Determining the requirement for threonine, as well as the availability of threonine from various food products will help us to develop better food recommendations for children.

Research Method This study will be carried out in a repeated measures design. Participants will be recruited and screened for eligibility. Six participants will be brought in for 6 testing visits with reference amino acid, where they will be randomized to a level of threonine intake. A further 3 visits will be carried out during which participants will be randomized to a level of threonine consumption derived from alternative proteins (casein, soy, peas) which is at a threshold below the requirement for threonine to determine availability.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 10 Y
* No history of chronic disease or metabolic disorders
* No food allergies
* No recent illness or antibiotic consumption
* Children with a normal, healthy, body weight (between 3rd and 85th percentiles for their age group for weight) (Dietitians of Canada, 2015)

Exclusion Criteria:

* Children under 6 years' old
* Children over 10 years' old
* Children with a history of disease or metabolic disorders
* Children with any food allergies
* Children taking prescription medication
* Children with a history of being underweight, overweight, or obese (Dietitians of Canada, 2015; Onis et al., 2007)

  o Below 3rd percentile for weight, Above 85th percentile for weight
* Female children who have commenced menstruation

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
13 Co2 production | 8 hours (1 study day)
  Urine and breath samples will be collected during the study day, to measure the rate of oxidation of tracer phenylalanine in the expired breath, and flux enrichment in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No